CLINICAL TRIAL: NCT02632747
Title: A Double-blind, Placebo Controlled, Cross-over Renal Mechanistic Trial to Assess the Effect of Adding Empagliflozin Versus Placebo on Renal Hyperfiltration on a Background of the Angiotensin Converting Enzyme Inhibitor (ACEi) Ramipril: BETWEEN Study
Brief Title: Empagliflozin and ACEi- Effects on Hyperfiltration: BETWEEN Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.100
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Obesity | interventions — empagliflozin; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sequence A (Experimental): Empagliflozin followed by a wash-out followed by empagliflozin matching placebo on a background of open label ramipril.
  Interventions: Drug: Empagliflozin; Drug: Placebo (matching empagliflozin); Drug: ramipril
- Sequence B (Experimental): Empagliflozin matching placebo followed a wash-out followed by empagliflozin on a background of open label ramipril.
  Interventions: Drug: Empagliflozin; Drug: Placebo (matching empagliflozin); Drug: ramipril

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin will be taken once daily
Drug: Placebo (matching empagliflozin) — Placebo will be taken once daily
Drug: ramipril — Ramipril will be taken once or twice daily

SUMMARY:
This is a randomized, double-blind, double-dummy, placebo-controlled, cross over design trial with empagliflozin compared to placebo that is added to open-label ramipril.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent.
* Male or female patients diagnosed with type 1 diabetes (T1D) at least 6 months prior to informed consent or type 2 diabetes (T2D) or non-diabetic obese patients.
* T1D patients must use and be willing of and be willing to continue throughout the duration of the trial either:
* multiple daily injections of insulin OR
* continuous sub-cutaneous insulin infusion of any insulin type, with at least 3 months experience
* For patients with T1D or T2D,HbA1c of 6.5 - 11%
* Age at least 18 years of age
* Body mass index of >=18.5 kg/m^2
* Estimated glomerular filtration rate greater than or equal to 60 ml/min/1.73m2
* Blood pressure greater than 90 /60 mmHg and less than or equal to 140 / 90 mmHg
* Use of a highly effective method of contraception.
* Further inclusion criteria apply

Exclusion criteria:

* For patients with T1D, treatment with an antihyperglycaemic agent within 3 months prior to visit 1
* occurrence of severe hypoglycaemia within 3 months prior to visit 1
* hypoglycaemic unawareness within 3 months prior to visit 1
* occurrence of diabetic ketoacidosis within 3 months of visit 1 and until visit 3 Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2019-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lytvyn Y, Kimura K, Peter N, Lai V, Tse J, Cham L, Perkins BA, Soleymanlou N, Cherney DZI. Renal and Vascular Effects of Combined SGLT2 and Angiotensin-Converting Enzyme Inhibition. Circulation. 2022 Aug 9;146(6):450-462. doi: 10.1161/CIRCULATIONAHA.122.059150. Epub 2022 Jul 11. PMID 35862082
- See also: Related Info — https://trials.boehringer-ingelheim.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blinded, placebo-controlled, crossover trial to compare the effect of empagliflozin versus placebo when added to ramipril on reducing glomerular hyperfiltration in patients with type 1 Diabetes mellitus (T1D), Type 2 Diabetes (T2D), or obesity.
Pre-assignment Details: Participants who successfully completed the 4 weeks open-label ramipril run-in period and meet all of the inclusion, and non of the exclusion criteria were randomized into the trial, with no stratification to one of two sequences.
Groups:
- Sequence A: 25 mg Empagliflozin / Placebo: During dosing Period 1, participants were administered 1 tablet of 25 milligram (mg) empagliflozin once daily as single oral dose for 4 weeks added to open-label Ramipril, where participants had been dose escalated from 1.25, 5, 7.5, or 10 mg, up to 10 mg ramipril or to their maximum tolerated dose. This was followed by a 4-week wash-out period with background treatment of open-label ramipril administered orally as capsule once or twice daily as prescribed by the investigator,and then followed by 4 weeks of dosing period 2 of 1 tablet matching placebo administered once daily as single oral dose added to open-label Ramipril.
- Sequence B: Placebo / 25 mg Empagliflozin: During dosing Period 1, participants were administered 1 tablet of matching placebo once daily as single oral dose for 4 weeks added to open-label Ramipril, where participants had been dose escalated from 1.25, 5, 7.5, or 10 mg, up to 10 mg ramipril or to their maximum tolerated dose. This was followed by a 4-week wash-out period with background treatment of open-label ramipril administered orally as capsule once or twice daily as prescribed by the investigator,and then followed by 4 weeks of dosing period 2 of 1 tablet of 25 mg empagliflozin administered once daily as single oral dose added to open-label Ramipril.
Period: Treatment Period 1
Arm/Group | Sequence A: 25 mg Empagliflozin / Placebo | Sequence B: Placebo / 25 mg Empagliflozin
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0
Period: Wash-out Period
Arm/Group | Sequence A: 25 mg Empagliflozin / Placebo | Sequence B: Placebo / 25 mg Empagliflozin
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2
Arm/Group | Sequence A: 25 mg Empagliflozin / Placebo | Sequence B: Placebo / 25 mg Empagliflozin
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS consists of all patients who were randomised, treated with at least one dose of empagliflozin/placebo and provided randomisation baseline (visit 8) and at least one post-randomisation glomerular filtration rate (GFR) measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A: 25 mg Empagliflozin / Placebo | Sequence B: Placebo / 25 mg Empagliflozin | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.5 (4.2) | 27.0 (5.0) | 26.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glomerular filtration rate (GFR) at baseline [Mean (Standard Deviation); unit: milliliter (mL) /minutes (min) /1.73m²] | 113.6 (9.4) | 115.7 (14.0) | 114.6 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate (GFR) Under Euglycaemic Conditions After 4 Weeks of Treatment With Either Empagliflozin Added to Ramipril or Placebo Added to Ramipril.
Description: Glomerular filtration rate (GFR) under euglycaemic conditions after 4 weeks of treatment with either empagliflozin added to ramipril or placebo added to ramipril.
  The pre-specified statistical analysis was not conducted, because data are too sparse in the subgroup of hyperfilterers.
Time Frame: At week 4 and at week 12
Population: Hyperfilterers: Patients before ramipril monotherapy with GFR ≥ 135 mL/min/1.73m², as measured at screening (visit 4).
Measure: Mean (Standard Deviation); unit: milliliter (mL) /minutes (min) /1.73m²
Groups:
- 25 mg Empagliflozin: Participants were administered 1 tablet of 25 milligram (mg) empagliflozin once daily as single oral dose, added to open-label Ramipril, where participants had been dose escalated from 1.25, 5, 7.5, or 10 mg, up to 10 mg Ramipril or to their maximum tolerated dose.
- Placebo: Participants were administered 1 tablet of matching placebo administered once daily as single oral dose, added to open-label Ramipril, where participants had been dose escalated from 1.25, 5, 7.5, or 10 mg, up to 10 mg Ramipril or to their maximum tolerated dose.
Arm/Group | 25 mg Empagliflozin | Placebo
Number analyzed (Participants) | 2 | 2
milliliter (mL) /minutes (min) /1.73m² | 124.0 (10.61) | 132.5 (7.78)

2. Secondary Outcome: Filtration Status (Glomerular Filtration Rate (GFR) < 120 mL/Min/1.73m², Yes/no) After 4 Weeks of Treatment With Either Empagliflozin Added to Ramipril or Placebo Added to Ramipril
Description: Filtration status (Glomerular Filtration Rate (GFR) < 120 mL/min/1.73m²) after 4 weeks of treatment with either empagliflozin added to ramipril or placebo added to ramipril. Filtration status is defined as whether a patient has normal Filtration status (GFR < mL/min/1.73m², "yes") or not (GFR ≥ mL/min/1.73m², "no").
  The pre-specified statistical analysis was not conducted, because data are too sparse in the subgroup of hyperfilterers.
Time Frame: At week 4 and at week 12.
Population: Hyperfilterers: Patients before ramipril monotherapy with GFR ≥ 135 mL/min/1.73m², as measured at screening (visit 4).
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg Empagliflozin | Placebo
Number analyzed (Participants) | 2 | 2
Participants
  Yes | 1 | 0
  No | 1 | 2

ADVERSE EVENTS:
Time Frame: From drug administration until 7 days after the last dose of treatment, up to 91 days.
Description: Treated Set (TS): All participants who were randomized and treated with at least one dose of double-blind study medication (empagliflozin, placebo).
Arm/Group | 25 mg Empagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/30
Other Adverse Events (participants affected / at risk) | 15/31 | 13/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg Empagliflozin (N=31) | Placebo (N=30)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Testicular rupture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg Empagliflozin (N=31) | Placebo (N=30)
Fatigue (General disorders) | 3 | 0
Thirst (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 3 | 7
Ketosis (Metabolism and nutrition disorders) | 6 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT02632747/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02632747/SAP_001.pdf